CLINICAL TRIAL: NCT04636684
Title: Prevalence and Significance of ATTR Aortic Valve Amyloidosis in Degenerative Aortic Stenosis
Acronym: RACAMYL
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: RC31/19/0446
Record Dates: First submitted 2020-11-13; First posted 2020-11-19 (Actual); Last update posted 2024-10-23 (Actual); Status verified 2024-10

CONDITIONS: Amyloidosis
Keywords: ATTR aortic valve amyloidosis
MeSH Terms: conditions — Amyloidosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- patients undergoing surgical valve replacement for degenerative aortic stenosis (Experimental)
  Interventions: Diagnostic Test: Proteomic analysis

INTERVENTIONS:
Diagnostic Test: Proteomic analysis — Proteomic analysis based on mass spectrometry on the sample of valve tissues.

SUMMARY:
Cardiac amyloidosis is a restrictive cardiomyopathy with a potentially severe prognosis that can be life-threatening. It is linked in the vast majority of cases to a light chain deposition of immunoglobulin or transthyretin. Although myocardial involvement is predominant, other locations are possible: the atrioventricular conduction system, coronary arteries and valve leaflets. In systematic histological analyzes, deposits of amyloidosis infiltrating the aortic valve have been reported with a frequency of up to 74% for degenerative RA. The nature of these deposits has never been established because the immunostaining carried out all remained negative, probably due to decalcification prior to cutting. Currently, these deposits are considered to be local degenerative phenomena without clinical repercussions. However, the use of bone scintigraphy has shown a high prevalence, between 14 and 16%, of ATTR cardiac amyloidosis in patients with severe RA. The diagnosis of ATTR amyloidosis has been proven histologically in a few patients. Sequencing of the TTR gene has shown that they are mainly wild forms. In fact, the prevalence of transthyretin mutations in our local cohort is 20%.

The objective of this study is to determine by proteomic analysis based on mass spectrometry, the prevalence of ATTR aortic valve amyloidosis in patients undergoing surgical valve replacement for degenerative aortic stenosis.

ELIGIBILITY:
Inclusion Criteria:

* Patient over 18 years old
* Degenerative aortic stenosis
* Aortic valve replacement surgery
* Signature of the informed consent form

Exclusion Criteria:

* Non-degenerative aortic stenosis: bicuspid, rheumatic disease, aortic regurgitation
* Persons under a system of legal protection for adults (guardianship, curatorship, etc.)
* Pregnant women

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-12-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
prevalence rate of valvular ATTR amyloidosis | 1 year
  calculation of the prevalence rate of valvular ATTR amyloidosis with its 95% confidence interval.

SECONDARY OUTCOMES:
Prevalence of ATTR myocardial amyloidosis revealed by bone scintigraphy | 1 year
  The prevalence of ATTR myocardial amyloidosis revealed by bone scintigraphy (HMDP scan) will be calculated
percentage of wild ATTR myocardial amyloidosis | 1 year
  The percentage of wild ATTR forms will be calculated
percentage of mutated ATTR myocardial amyloidosis | 1 year
  The percentage of mutated ATTR forms will be calculated
Prevalence of types of amyloidosis other than ATTR | 1 year
  The prevalence of types of amyloidosis other than ATTR will be calculated

CONTACTS AND LOCATIONS:
Overall Officials: Magali COLOMBAT, MD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- university hospital center Toulouse, Toulouse, France